CLINICAL TRIAL: NCT05140408
Title: Efficiency of the Imaging Strategy for the Management of Pneumonia in the Emergency Department
Brief Title: Efficiency of the Imaging Strategy for the Management of Pneumonia
Acronym: EFFI-PNEUMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8129
Record Dates: First submitted 2021-10-13; First posted 2021-12-01 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia
Keywords: Pneumonia; Emergency; Imaging strategy; pneumopathy; Hemodynamic complications; Antibiotic therapy
MeSH Terms: conditions — Pneumonia; Emergencies; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For patients with suspected pneumonia presenting to the emergency room, the imaging strategy most often involves a frontal and lateral chest x-ray despite poor diagnostic input. Indeed, the radiography is not very sensitive and specific for the diagnosis of pneumopathy compared to the scanner. However, the scanner remains the gold standard, the major constraint of which concerns the irradiation to which the patient is exposed. The new scanners allow ultra-low-dose scans with better sensitivity than standard radiography with an equivalent dose of radiation. In addition, the ultra-low-dose scanner helps prevent diagnostic errors and unintended treatments. A low-dose CT scan for suspected pneumonia has been possible in the Strasbourg emergency department since March 2019. The investigators therefore hypothesize that a diagnostic strategy involving the performance of a low dose CT scan in the event of suspicion of pneumopathy in the emergency room makes it possible to improve the adequacy of the diagnosis made by the initial imaging examination and the diagnosis on discharge from hospitalization, to reduce respiratory or hemodynamic complications and to reduce the prescription of antibiotic therapy that is not suitable for the patient. course of the imaging result validated by a panel of emergency physicians and infectious disease specialists based on medical records in accordance with the recommendations.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Emergency consultant subject with a final diagnosis of pneumonia, diagnostic code J18 and J15 with imaging: standard radiography or low dose scanner from 03/01/2019 to 02/29/2020
* Subject not having expressed their opposition, after information, to the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Absence of emergency imaging
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject consulting the emergency department and had a final diagnosis of pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 2240 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Study of the imaging strategy for the management of patients with pneumonia in emergency departments | Files analysed retrospectively from March 01, 2019 to February 29, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Accueil des Urgences - Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Kepka S, Zarca K, Ohana M, Hoffbeck L, Heimann C, Borgne PL, Severac F, Muller J, Sauleau EA, Bilbault P, Zaleski ID. Cost effectiveness of imaging strategies in the emergency department for the diagnostic workup of community-acquired pneumonia: a real-life retrospective study. Health Econ Rev. 2025 May 20;15(1):41. doi: 10.1186/s13561-025-00625-8. PMID 40392398